CLINICAL TRIAL: NCT02639598
Title: Flunarizine Versus Topiramate for Chronic Migraine Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Deputy Head, Neurological Institute, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-04-046B
Record Dates: First submitted 2015-12-16; First posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Migraine
Keywords: chronic migraine; prophylaxis; flunarizine; topiramate
MeSH Terms: interventions — Flunarizine; Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- flunarizine (Experimental): This study consisted of two periods: a prospective baseline screening period lasting up to 2 weeks (week -2 to week 0, T0), and a treatment period lasting 8 weeks after enrollment (weeks 0-8, T1-T4).
  The treatment phase consisted of a 2-week titration period (T1) and a 6-week maintenance period (T2-T4). During the titration period, subjects were given 5 mg/day flunarizine once daily in the first week, followed by 10 mg/day flunarizine in divided doses (twice daily) in the second week. When subjects could not tolerate this target dose, the initial dose was continued through T4.
  Interventions: Drug: Flunarizine
- topiramate (Active Comparator): This study consisted of two periods: a prospective baseline screening period lasting up to 2 weeks (week -2 to week 0, T0), and a treatment period lasting 8 weeks after enrollment (weeks 0-8, T1-T4).
  The treatment phase consisted of a 2-week titration period (T1) and a 6-week maintenance period (T2-T4). During the titration period, subjects were given 25 mg/day topiramate once daily in the first week, followed by 50 mg/day topiramate in divided doses (twice daily) in the second week. When subjects could not tolerate this target dose, the initial dose was continued through T4.
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Flunarizine — as in "arm descriptions"
  Other Names: sibelium
  Arms: flunarizine
Drug: Topiramate — as in "arm descriptions"
  Other Names: topamax
  Arms: topiramate

SUMMARY:
Chronic migraine (CM) is a prevalent and devastating disorder with limited therapeutic options. This study explored the efficacy of 10 mg/day flunarizine for CM prophylaxis as compared with 50 mg/day topiramate.

DETAILED DESCRIPTION:
Chronic migraine (CM) is a prevalent and devastating disorder with limited therapeutic options. This study explored the efficacy of 10 mg/day flunarizine for CM prophylaxis as compared with 50 mg/day topiramate.

We conducted a prospective, randomized, open-label, blinded-endpoint (PROBE) trial. Patients with CM were randomized (1:1) to flunarizine and topiramate treatment groups.

This study consisted of two periods: a prospective baseline screening period lasting up to 2 weeks (week -2 to week 0, T0), and a treatment period lasting 8 weeks after enrollment (weeks 0-8, T1-T4).

The treatment phase consisted of a 2-week titration period (T1) and a 6-week maintenance period (T2-T4). During the titration period, subjects were given 25 mg/day topiramate or 5 mg/day flunarizine once daily in the first week, followed by 50 mg/day topiramate or 10 mg/day flunarizine in divided doses (twice daily) in the second week. When subjects could not tolerate this target dose, the initial dose was continued through T4.

Patients were followed per 2 weeks at the Headache Clinic. At each visit, diaries were collected and directed to the outcome evaluators, who were blinded to the patients' treatment.

The primary outcomes assessed were the reductions in the total numbers of headache days and migraine days after 8 weeks of treatment (weeks 7 to 8 vs. weeks -2 to 0). Secondary outcomes were reductions in the numbers of days of acute abortive medication intake and acute abortive medication tablets taken, and the 50% responder rate.

ELIGIBILITY:
Inclusion Criteria:

* ICHD-IIR criteria for CM (as reported by the patient)
* Experienced ≥7 days of headache lasting ≥30 min during T0 (-2 week to 0 week).
* On ≥4 of these days, subjects were required to have experienced migrainous headache
* Prophylaxis-naïve (i.e., patients could not receive any preventive medications)
* With and without medication overuse

Exclusion Criteria:

* Headache type other than CM
* Migraine onset after the age of 50 years
* CM onset after the age of 60 years
* Previous history of migraine prophylaxis before enrollment
* Pregnancy or nursing status
* History of hepatic or renal disorder, nephrolithiasis or other severe systemic disease
* Severe depression (BDI score ≥ 30 at visit 1)
* Conditions incompatible with MRI, such as claustrophobia or metallic or electric implants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
reduction of total number of headache days (by diary log) | week 7 to 8 after treatment (T4) compared to week -2 to 0 before treatment (T0)
  Patients were followed per 2 weeks at the Headache Clinic. At each visit, diaries were collected, and information within the diary was used for outcome measurement.
reduction of number of migraine days (by diary log) | week 7 to 8 after treatment (T4) compared to week -2 to 0 before treatment (T0)
  Patients were followed per 2 weeks at the Headache Clinic. At each visit, diaries were collected, and information within the diary was used for outcome measurement.

SECONDARY OUTCOMES:
reduction of number of days of acute abortive medication intake (by diary log) | week 7 to 8 after treatment (T4) compared to week -2 to 0 before treatment (T0)
  Patients were followed per 2 weeks at the Headache Clinic. At each visit, diaries were collected, and information within the diary was used for outcome measurement.
reduction of number of acute abortive medication tablets taken (by diary log) | week 7 to 8 after treatment (T4) compared to week -2 to 0 before treatment (T0)
  Patients were followed per 2 weeks at the Headache Clinic. At each visit, diaries were collected, and information within the diary was used for outcome measurement.
fifty percent responder rate (by diary log) | week 7 to 8 after treatment (T4) compared to week -2 to 0 before treatment (T0)
  Patients were followed per 2 weeks at the Headache Clinic. At each visit, diaries were collected, and information within the diary was used for outcome measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Shuu-Jiun Wang, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis D, Ashwal S, Hershey A, Hirtz D, Yonker M, Silberstein S; American Academy of Neurology Quality Standards Subcommittee; Practice Committee of the Child Neurology Society. Practice parameter: pharmacological treatment of migraine headache in children and adolescents [RETIRED]: report of the American Academy of Neurology Quality Standards Subcommittee and the Practice Committee of the Child Neurology Society. Neurology. 2004 Dec 28;63(12):2215-24. doi: 10.1212/01.wnl.0000147332.41993.90. PMID 15623677
- [Background] Evers S, Afra J, Frese A, Goadsby PJ, Linde M, May A, Sandor PS; European Federation of Neurological Societies. EFNS guideline on the drug treatment of migraine--revised report of an EFNS task force. Eur J Neurol. 2009 Sep;16(9):968-81. doi: 10.1111/j.1468-1331.2009.02748.x. PMID 19708964
- [Background] Pringsheim T, Davenport W, Mackie G, Worthington I, Aube M, Christie SN, Gladstone J, Becker WJ; Canadian Headache Society Prophylactic Guidelines Development Group. Canadian Headache Society guideline for migraine prophylaxis. Can J Neurol Sci. 2012 Mar;39(2 Suppl 2):S1-59. PMID 22683887
- [Background] Treatment Guideline Subcommittee of the Taiwan Headache Society. [Treatment guidelines for preventive treatment of migraine]. Acta Neurol Taiwan. 2008 Jun;17(2):132-48. Chinese. PMID 18686655
- [Result] Silvestrini M, Bartolini M, Coccia M, Baruffaldi R, Taffi R, Provinciali L. Topiramate in the treatment of chronic migraine. Cephalalgia. 2003 Oct;23(8):820-4. doi: 10.1046/j.1468-2982.2003.00592.x. PMID 14510929
- [Result] Bartolini M, Silvestrini M, Taffi R, Lanciotti C, Luconi R, Capecci M, Provinciali L. Efficacy of topiramate and valproate in chronic migraine. Clin Neuropharmacol. 2005 Nov-Dec;28(6):277-9. doi: 10.1097/01.wnf.0000192136.46145.44. PMID 16340383
- [Result] Diener HC, Bussone G, Van Oene JC, Lahaye M, Schwalen S, Goadsby PJ; TOPMAT-MIG-201(TOP-CHROME) Study Group. Topiramate reduces headache days in chronic migraine: a randomized, double-blind, placebo-controlled study. Cephalalgia. 2007 Jul;27(7):814-23. doi: 10.1111/j.1468-2982.2007.01326.x. Epub 2007 Apr 18. PMID 17441971
- [Result] Silberstein SD, Lipton RB, Dodick DW, Freitag FG, Ramadan N, Mathew N, Brandes JL, Bigal M, Saper J, Ascher S, Jordan DM, Greenberg SJ, Hulihan J; Topiramate Chronic Migraine Study Group. Efficacy and safety of topiramate for the treatment of chronic migraine: a randomized, double-blind, placebo-controlled trial. Headache. 2007 Feb;47(2):170-80. doi: 10.1111/j.1526-4610.2006.00684.x. PMID 17300356
- [Result] Silberstein S, Lipton R, Dodick D, Freitag F, Mathew N, Brandes J, Bigal M, Ascher S, Morein J, Wright P, Greenberg S, Hulihan J. Topiramate treatment of chronic migraine: a randomized, placebo-controlled trial of quality of life and other efficacy measures. Headache. 2009 Sep;49(8):1153-62. doi: 10.1111/j.1526-4610.2009.01508.x. PMID 19719543
- [Result] Martinez-Lage JM. Flunarizine (Sibelium) in the prophylaxis of migraine. An open, long-term, multicenter trial. Cephalalgia. 1988;8 Suppl 8:15-20. doi: 10.1177/03331024880080S804. PMID 3052850
- [Result] Visudtibhan A, Lusawat A, Chiemchanya S, Visudhiphan P. Flunarizine for prophylactic treatment of childhood migraine. J Med Assoc Thai. 2004 Dec;87(12):1466-70. PMID 15822542
- [Result] Li HL, Kwan P, Leung H, Yu E, Tsoi TH, Hui AC, Sheng B, Lau KK. Topiramate for migraine prophylaxis among Chinese population. Headache. 2007 Apr;47(4):616-9. doi: 10.1111/j.1526-4610.2007.00763_3.x. PMID 17445114